CLINICAL TRIAL: NCT07315893
Title: Endoscopic Full Thickness Suturing of Mucosal, Submucosal and Perforation Defects Using Su2ura® GI System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anchora Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANC-201
Record Dates: First submitted 2025-12-21; First posted 2026-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Endoscopic Mucosal Resection; Endoscopic Submucosal Dissection (ESD)
Keywords: endoscopic mucosal resection (EMR); endoscopic submucosal dissection (ESD); a gastric neoplastic lesion
MeSH Terms: interventions — Physical Examination; Vital Signs; Gastroscopy; Pain Measurement

STUDY DESIGN:
Intervention Model Description: All participants will undergo endoscopic suturing using a Su2ura® GI System following the ESD or EMR procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Su2ura® GI System-study device group (Experimental): All participants will undergo endoscopic suturing using a Su2ura® GI System following the ESD or EMR procedure.
  Interventions: Device: Su2ura® GI system; Diagnostic Test: Physical Examination; Diagnostic Test: Vital Signs; Diagnostic Test: Blood Test-Hematology; Diagnostic Test: Blood Test-Biochemistry; Diagnostic Test: Urine Pregnancy Test; Diagnostic Test: Gastroscopy; Diagnostic Test: Health-related quality of life (HR-QoL); Diagnostic Test: Visual Analogue Scale (VAS)

INTERVENTIONS:
Device: Su2ura® GI system — The Su2ura® GI handle is used to control tissue grasping, anchor deployment, and suture placement, enabling controlled full-thickness tissue approximation through sequential deployment of T-Tag Anchors in a predefined suturing pattern.
Diagnostic Test: Physical Examination — The patient will undergo a standard physical examination by an authorized physician. The physician's evaluation will include diagnosis and documentation of any significant clinical abnormalities or diseases.
Diagnostic Test: Vital Signs — Vital signs include blood pressure, pulse, temperature, body weight and height, BMI.
Diagnostic Test: Blood Test-Hematology — All subjects will undergo Hematology blood tests. Blood Hematology and Biochemistry will include standard of care measurements. 5 ml of blood (equals to 1 spoon) will be taken for each test.
Diagnostic Test: Blood Test-Biochemistry — All subjects will undergo Biochemistry blood tests. Blood Hematology and Biochemistry will include standard of care measurements. 5 ml of blood (equals to 1 spoon) will be taken for each test.
Diagnostic Test: Urine Pregnancy Test — Women with child-bearing potential will undergo a urine pregnancy test during the screening visit.
Diagnostic Test: Gastroscopy — During visit 4 (Day 28 ± 2 days after procedure) a gastroscopy examination will be performed, to negate local recurrence. The examination will be performed as accepted, with a gastroscope with an NBI/BLI optical filter. Biopsies will be sampled as needed, at a gastroenterologist's discretion.
Diagnostic Test: Health-related quality of life (HR-QoL) — A questionnaire assessing patient-reported satisfaction and function.
Diagnostic Test: Visual Analogue Scale (VAS) — A validated, subjective measure measuring acute and chronic pain.

SUMMARY:
The objective of this clinical study is to assess the safety of the Su2ura® GI system when used for endoscopic suturing and soft-tissue approximation in patients referred for endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of gastric neoplastic lesions.

The main questions it aims to answer are:

1. Percentage of patients with incomplete closure.
2. Percentage of patients bleeding at closure site within 28 days from procedure.
3. Percentage of patients with infection at closure site within 28 days from procedure.
4. Percentage of patients with leakage within 72 hours from procedure.
5. Serious Adverse Device Effects (SADE) within 28 days from procedure.
6. Overall rates of Adverse Device Effect within 28 days from procedure.

Study includes 6 visits: Screening, Baseline/Surgery, Discharge and 4 weeks, 3 months and 6 months post-surgery. The actual point of enrollment for each subject is considered the day of surgery. Total study duration is up to 6.5 months.

The patient will be admitted to the medical center on the day of the procedure or one day prior for preoperative preparation. Following tissue resection using one of the methods (ESD or EMR), suturing will be performed using the Su2ura® GI system.

Postoperatively, the patient will be transferred to the recovery area and then to the surgical ward for standard monitoring, with an expected one-night postoperative stay and discharge the following day.

Study follow-up visits will take place 4 weeks, 3 and 6 months post surgery.

DETAILED DESCRIPTION:
This study will be performed in accordance with the design and specific provisions of this protocol, in accordance with the ethical principles that have their origin in the Declaration of Helsinki, that are consistent with Good Clinical Practice (GCP), Title 21 of the Code of Federal Regulations (21 CFR), part 812 (Investigational Device Exemptions), and the applicable regulatory requirements.

The study will be a prospective, single-center, open study, to evaluate the efficacy and safety of the Su2ura® GI System.

The study will be performed at the Tel Aviv Sourasky Medical Center, Israel. Up to 25 patients will be recruited to the study.

Following resection of the lesion using either endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD), the procedure involves endoscopic insertion of the Su2ura® GI system through the gastroscope working channel, followed by tissue grasping and approximation using sequential deployment of T-Tag Anchors in a predefined suturing pattern. Full-thickness anchors are placed in a controlled manner to achieve safe and effective tissue approximation, after which the suture is secured using the Su2ura® Knot device.

Postoperatively, the patient will be transferred to the recovery area and then to the surgical ward for standard monitoring, with an expected one-night postoperative stay and discharge the following day.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patient is able to provide informed consent .
3. Body mass index (BMI) 20-40 kg/m2
4. Patient is referred for endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of a gastric neoplastic lesion
5. Candidate for endoscopic defect closure based on the operating's endoscopist assessment.

Exclusion Criteria:

1. Patient with severe comorbidities likely to limit survival to less than 2 years.
2. Patients with INR>1.5
3. Patients with PLT< 150
4. Patient with known collagen or connective tissue disorders (e.g. scleroderma, marfan syndrome) .
5. Pregnant women or those intending to become pregnant during the study period
6. Patient with ascites on physical examination or CT scan.
7. Patient with varices.
8. Patient on peritoneal dialysis.
9. Patient with wound-healing disorders.
10. Patient with significant coagulation disorders or those requiring anti thrombotic or anticoagulation treatment other than aspirin .
11. Patient with autoimmune disorder requiring more than 10 mg of corticosteroid daily .
12. Patients in need of immunomodulatory therapy.
13. Immunocompromised patients (e.g., HIV/AIDS, organ transplant, chemo- or radiation therapy 6 months prior to recruitment).
14. Patient in need of concomitant surgical procedures other than those permitted in the protocol.
15. Non-compliance with the study protocol.
16. Patient requests to exist the study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients with incomplete closure. | Up to 28 days
  Percentage of patients with incomplete closure.
Patients bleeding at closure site. | Up to 28 days
  Percentage of patients bleeding at closure site within 28 days from procedure.
Patients with infection at closure site. | Up to 28 days
  Percentage of patients with infection at closure site within 28 days from procedure.
Patients with leakage. | Up to 72 hours
  Percentage of patients with leakage within 72 hours from procedure.
Serious Adverse Device Effects (SADE) | Up to 28 days
  Serious Adverse Device Effects (SADE) within 28 days from procedure.
Overall rates of Adverse Device Effect | Up to 28 days
  Overall rates of Adverse Device Effect within 28 days from procedure.

SECONDARY OUTCOMES:
Overall rates of Serious Adverse Events | Up to 180 days
  Overall rates of Serious Adverse Events will be recorded up to 180 days following the procedure.
Serious Adverse Device Effects | Up to 90 days
  Serious Adverse Device Effects (SADE) will be evaluated endoscopically at 2-14 and 90 days.
Evidence of a Leak | Up to 30 days
  Clinical, radiologic or endoscopic evidence of a Leak within 30 days
Patient Quality of Life | Up to 180 days
  Patient quality of life will be assessed by validated Health-Related Quality of Life Scale questionnaire.
  The questionnaire includes several measures of perceived health status. The primary overall outcome is the Unhealthy Days Score, calculated as the sum of the number of days of poor physical health and poor mental health during the past 30 days. The score ranges from 0 to 30 days, with higher scores indicating worse health status and lower scores indicating better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Ichilov, Tel Aviv, Israel